CLINICAL TRIAL: NCT05089760
Title: Microbiology, Antimicrobial Resistance and Outcomes of Neonatal Sepsis in Chinese Neonatal Intensive Care Units
Brief Title: Microbiology, Antimicrobial Resistance and Outcomes of Neonatal Sepsis in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Chinese Neonatal Network (Other)
Responsible Party: Sponsor
Other Study IDs: MAROC-ChiNICU
Record Dates: First submitted 2021-09-06; First posted 2021-10-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Antimicrobial Resistance; Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with bacteria sepsis: Infants diagnosed with culture-proven sepsis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a prospective observational cohort study. The purpose of the study was to compare the incidence of mortality, complications, and other outcomes between infants with multi-resistant bacteria sepsis and infants with sepsis caused by non-multi-resistant bacteria, and compare the incidence of complications and other outcomes between infants with sepsis-related death and infants who survive.

SUMMARY:
Neonatal sepsis remains one of the most important cause of mortality and morbidities in China. This study will establish a prospective registral cohort of all infants with culture-proven neonatal sepsis in Chinese NICUs participating in the Chinese Neonatal Network (CHNN). The microbiology, antimicrobial resistance patterns and neonatal outcomes will be described in detail for this cohort.

DETAILED DESCRIPTION:
All infants with culture-proven sepsis in NICUs of CHNN will be enrolled in the study. Detailed data on microbiology, resistance pattern, neonatal mortality and morbidities will be collected and described. Risk factors for multi-resistant bacteria infections and for sepsis-related mortality will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to CHNN NICUs from 2022.1.1 to 2023.12.31
* Diagnosed with culture-proven sepsis

Exclusion Criteria:

* None

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates diagnosed with culture-proven sepsis and admitted to CHNN NICUs from 2022.1.1 to 2023.12.31
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | About 3 months from admission to discharge or death
  Incidence of death during the study period

SECONDARY OUTCOMES:
Sepsis-related mortality (within 7 days of sepsis) | About 3 months from admission to discharge or death
  Incidence of death within 7 days after sepsis
Incidence of multiorgan dysfunction | About 3 months from admission to discharge or death
  Propertion of infants who occur multiorgan dysfunction
Incidence of septic shock | About 3 months from admission to discharge or death
  Propertion of infants who occur septic shock
Incidence of respiratory failure | About 3 months from admission to discharge or death
  Propertion of infants who occur respiratory failure
Incidence of disseminated intravascular coagulation (DIC) | About 3 months from admission to discharge or death
  Propertion of infants who occur DIC
Incidence of renal failure | About 3 months from admission to discharge or death
  Propertion of infants who accur renal failure
Incidence of meningitis | About 3 months from admission to discharge or death
  Propertion of infants who accur meningitis
Incidence of necrotizing enterocolitis | About 3 months from admission to discharge or death
  Propertion of infants who accur necrotizing enterocolitis
Incidence of brain injury | About 3 months from admission to discharge or death
  Propertion of infants who accur brain injury
Length of hospital stay | About 3 months from admission to discharge or death
  Days of hospitalization
Length of antibiotic treatment | About 3 months from admission to discharge or death
  Days of antibiotic treatment
Type and quantity of transfusion | About 3 months from admission to discharge or death
  Which kind and how much (ml) of blood product was used during the study

CONTACTS AND LOCATIONS:
Overall Officials: Yun Cao, Ph.D, M.D., Principal Investigator — Children's Hospital of Fudan University, Shanghai, China